CLINICAL TRIAL: NCT00553540
Title: A Randomized Prospective Study to Evaluate the Effectiveness of Orthopedic Spinal Supports in the Treatment of Low Back Pain
Brief Title: Study to Evaluate the Effectiveness of Orthopedic Spinal Supports in the Treatment of Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cleveland Clinic Florida (Other)
Collaborators: Integral Orthopedics Inc. (Industry)
Responsible Party: Sponsor
Organization: The Cleveland Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IOI
Record Dates: First submitted 2007-11-02; First posted 2007-11-05 (Estimated); Results first posted 2019-11-25 (Actual); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Low Back Pain
Keywords: backache; low backpain; sciatica
MeSH Terms: conditions — Low Back Pain; Back Pain; Sciatica

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control Group (No Intervention): Patients in this group will receive physical therapy and posture education for low back pain
- Test Group (Active Comparator): Patients in this group will receive spinal / back supports in addition to physical therapy and posture education for low back pain
  Interventions: Device: Back supports

INTERVENTIONS:
Device: Back supports — The spinal / back supports are made of polymer shield covered by fabric and foam to be used externally to relieve back pain and offer spinal support. They are to be placed in the chair used in workstation related jobs.
  Other Names: Moller Back Support System
  Arms: Test Group

SUMMARY:
The purpose of this study is to determine whether orthopedic spinal supports are effective in the treatment of low back pain.

DETAILED DESCRIPTION:
Back pain is a common and expensive medical condition. Although rarely life-threatening, back disorders are a major cause of pain, disability, and social cost affecting the quality of life in most patients. Although primary care providers routinely treat back pain, little is known about how often primary care providers manage occupation-related symptoms and how outcomes compare with other treatment modalities. Treatment outcomes utilizing a non-operative treatment paradigm have not been adequately studied. This paradigm consists of treating patients sequentially with analgesics, physical therapy, use of back supports, caudal epidural steroid injections, or surgical referral. The use of spinal supports as a complimentary treatment along with physical therapy and posture education is promising.

ELIGIBILITY:
Inclusion Criteria:

* Patients must present with clinical symptoms of low back pain and evaluated by the study physician
* Visual Analog Score (VAS) for Pain >6 in response to the following question: Circle one number (from 0 = no pain to 10 = worst pain) "How would you rate the worst pain you experienced in last week."
* Patients must have x-ray and or an MRI film for diagnostic evaluation based on physician judgment.
* Age >18; both male and female
* Pain duration >3 months

Exclusion Criteria:

* Prior use of opioids, physical therapy, epidural injections for back pain or ongoing chiropractor care and or acupuncture treatment
* Moderate to severe arthritis of the spine/ knee or hip that might severely compromise ambulation and or posture
* Patients with diagnosed lumbar canal stenosis
* Serious concomitant medical illness (i.e., heart disease)
* Obese patients (twice the width of the Moller Orthopedic Back Support)
* Patients with moderate to severe scoliosis
* Past or present existence of a movement disorder, e.g., Parkinsonism, or any neurological disease that might affect ambulation and or postural changes History of osteoporosis
* Severe psychiatric disorder
* Prior spine surgery
* Multiple vertebral compression fractures with kyphosis
* Past or present workmen's compensation claim, SSI disability, or ongoing litigation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2006-10; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vinod K Podichetty, MD,MS, Study Director — Cleveland Clinic Florida; David Westerdahl, MD, Principal Investigator — Cleveland Clinic Florida
Locations (1):
- Cleveland Clinic Florida, Weston, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Andersson GBJ. The epidemiology of spinal disorders. In: Frymoyer JW, Ducker TB, Hadler NM, et al, eds. The Adult Spine: Principles and Practice. Philadelphia: Lippincott-Raven, 1997:93-141.
- [Background] Leboeuf-Yde C, Lauritsen JM. The prevalence of low back pain in the literature. A structured review of 26 Nordic studies from 1954 to 1993. Spine (Phila Pa 1976). 1995 Oct 1;20(19):2112-8. doi: 10.1097/00007632-199510000-00009. PMID 8588168
- [Background] Frymoyer JW, Durett CL. The economics of spinal disorders. In: Frymoyer JW, Ducker TB, Hadler NM, et al, eds. The Adult Spine: Principles and Practice. Philadelphia: Lippincott-Raven, 1997:143-150.
- [Background] Hart LG, Deyo RA, Cherkin DC. Physician office visits for low back pain. Frequency, clinical evaluation, and treatment patterns from a U.S. national survey. Spine (Phila Pa 1976). 1995 Jan 1;20(1):11-9. doi: 10.1097/00007632-199501000-00003. PMID 7709270
- [Background] Coste J, Delecoeuillerie G, Cohen de Lara A, Le Parc JM, Paolaggi JB. Clinical course and prognostic factors in acute low back pain: an inception cohort study in primary care practice. BMJ. 1994 Feb 26;308(6928):577-80. doi: 10.1136/bmj.308.6928.577. PMID 8148683
- [Background] Deyo RA, Phillips WR. Low back pain. A primary care challenge. Spine (Phila Pa 1976). 1996 Dec 15;21(24):2826-32. doi: 10.1097/00007632-199612150-00003. PMID 9112706
- [Background] Carey TS, Garrett JM, Jackman A, Hadler N. Recurrence and care seeking after acute back pain: results of a long-term follow-up study. North Carolina Back Pain Project. Med Care. 1999 Feb;37(2):157-64. doi: 10.1097/00005650-199902000-00006. PMID 10024120
- [Background] Bernard BP. Introduction. In: Bernard BP, ed. Musculoskeletal Disorders and Workplace Factors. Cincinnati: National Institute for Occupational Safety and Health, Centers for Disease Control, U.S. Department of Health and Human Services, 1997.
- [Background] Murphy PL, Volinn E. Is occupational low back pain on the rise? Spine (Phila Pa 1976). 1999 Apr 1;24(7):691-7. doi: 10.1097/00007632-199904010-00015. PMID 10209800
- [Background] van Tulder MW, Koes BW, Bouter LM. Conservative treatment of acute and chronic nonspecific low back pain. A systematic review of randomized controlled trials of the most common interventions. Spine (Phila Pa 1976). 1997 Sep 15;22(18):2128-56. doi: 10.1097/00007632-199709150-00012. PMID 9322325
- [Derived] Podichetty VK, Varley ES. Spinal supports and physical therapy in patients with low back pain: a case series. BMJ Case Rep. 2009;2009:bcr07.2008.0405. doi: 10.1136/bcr.07.2008.0405. Epub 2009 Apr 23. PMID 21686825

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control Group | Test Group
Started | 25 | 25
Completed | 23 | 20
Not Completed | 2 | 5
Not completed — discharged after first visit | 2 | 5

BASELINE CHARACTERISTICS:
Population: A total of 43 participants for whom baseline characteristics were measured.
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Test Group | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: We did not have the age for several participants and were regarded as missing values when running the data in SPSS
  years
    number analyzed (Participants) | 23 | 20 | 43
    (all) | 48.48 (9.462) | 42.95 (11.781) | 45.61 (10.98)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: the analyzed number of participants is different because, complete data was only collected for the numbers given. The other seven had incomplete data
  Participants
    number analyzed (Participants) | 23 | 20 | 43
    Female | 13 | 14 | 27
    Male | 10 | 6 | 16
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] — Population: The analyzed number of participants is different because, complete data was only collected for the numbers given. The other seven had incomplete data
  kg/m^2
    number analyzed (Participants) | 23 | 20 | 43
    (all) | 28.326 (6.498) | 28.686 (5.997) | 28.49 (6)

OUTCOME MEASURES:

1. Primary Outcome: Change in Low Back Pain
Description: numeric pain scale was used to determine pain at 1 week intervals starting from week 1 to week 24. Pain scores were determined by the numeric pain score of 1 to 10 (1 being the least painful to 10 being the highest level of pain) then summed up and averaged at 24 time points at 1 week intervals starting from week 1 to week 24.
Time Frame: 6 months
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Control Group | Test Group
Number analyzed (Participants) | 23 | 20
units on a scale | 2.58 [1 to 10] | 1.80 [1 to 10]

ADVERSE EVENTS:
Time Frame: adverse events were not monitored or assessed
Description: adverse events were not monitored or assessed
Arm/Group | Control Group | Test Group
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No